CLINICAL TRIAL: NCT03798938
Title: Effects of Plant-Based Diet on Peripheral Arterial Disease
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Vascular Institute of Texas (Other)
Responsible Party: Sponsor
Other Study IDs: 01012019
Record Dates: First submitted 2019-01-07; First posted 2019-01-10 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Diet, Plant-Based

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: plant-based diet — subjects will be placed in plant-based diet and the effect of plant-based diet to the endothelial function will be monitored

SUMMARY:
Cardiovascular disease (CVD), a condition predominantly caused by atherosclerosis, is the leading cause of morbidity and mortality in the investigator's society. Peripheral arterial disease (PAD), a subset of CVD, occurs when the atherosclerosis progresses to compromise the lower extremity circulation resulting in ischemic symptoms. Although atherosclerosis has been generally regarded as a disease of developed or affluent countries, recent evidence showed a progressive rise in the prevalence of CVD in developing countries where an epidemiological shift of disease prevalence patterns from infectious illnesses to atherosclerotic disease has occurred. Management of CVD, particularly with an emphasis of disease prevention, will undoubtedly play an increasing vital role in the health care system around the world.

Endothelial dysfunction, as reflected by the impaired arterial vasodilatory capacity, represents one of the pathogenic mechanisms linking atherosclerosis and cardiovascular mortality. The ability of arteries to dilate in response to stimuli is a significant indicator of underlying vascular endothelial function and associated CVD. Factors modulating vasodilatory response include the release of vasoactive compounds such as nitric oxide (NO) from the endothelium and vascular compliance. In healthy individuals, a major mechanism responsible for vasodilation is the hyperemic-stimulated release of NO from the endothelium, resulting in vascular smooth muscle relaxation with subsequent vasodilation.

Vascular endothelial function can be assessed using a non-invasive technique to determine brachial artery reactivity whereby a high-resolution ultrasound is used to measure changes in brachial artery diameter to endogenous production of endothelium-derived NO via flow-mediated dilation (FMD). Therefore, reduced FMD has been described as a reliable indicator of vascular endothelial dysfunction as well as presence of underlying CVD risk factors and related diseases. Recent studies have similarly shown that arterial pulse-wave velocity (PWV), which is a non-invasive evaluation of arterial stiffness, is a reliable indicator of vascular function. While numerous studies have documented the benefit of dietary intervention in the reduction of CVD related sequelae, limited data is available regarding whether the beneficial effect of dietary intervention are reflected in vascular endothelial function. The present study was therefore conducted to assess the effects of plant-based diet (PBD) on vascular endothelial function as assessed by FMD and PWV in patients with peripheral arterial disease (PAD).

DETAILED DESCRIPTION:
Patients with peripheral arterial disease (PAD) will be included in the study. Inclusion criteria for PAD included an ankle brachial index (ABI) of 0.90 or less at baseline. Those with an ABI greater than 0.90 at baseline were eligible if a non-invasive vascular ultrasound demonstrated PAD, lower extremity angiography showed arterial stenosis of 70% or greater, or medical records documented prior revascularization of lower extremities.9 Additionally, subjects must be willing and able to maintain an on-line food journal using smartphone-based dietary apps. Once enrolled, all participants underwent baseline evaluation, after which they were enrolled in either dietary advice for plant-based diet (PBD group) or no specific dietary advice (control group). The dietary intervention was continued for four months, at the end of which a follow up evaluation was performed.

ELIGIBILITY:
Inclusion Criteria:

* peripheral arterial disease

Exclusion Criteria:

* none

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: peripheral arterial disease as defined by an ankle brachial index (ABI) of 0.90 or less at baseline. Those with an ABI greater than 0.90 at baseline will be eligible if a non-invasive vascular ultrasound demonstrated PAD, lower extremity angiography showed arterial stenosis of 70% or greater, or medical records documented prior revascularization of lower extremities
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-01-10 (Estimated); Primary Completion 2019-06-10 (Estimated); Study Completion 2019-10-10 (Estimated)

PRIMARY OUTCOMES:
endothelial function | 10 minutes
  brachial artery reactivity test, flow-mediated vasodilation

CONTACTS AND LOCATIONS:
Locations (1):
- University Vascular Associates, Alhambra, California, United States

IPD SHARING:
Plan to Share IPD: No